CLINICAL TRIAL: NCT03445195
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of Intravenous Sulbactam-ETX2514 in the Treatment of Hospitalized Adults With Complicated Urinary Tract Infections, Including Acute Pyelonephritis
Brief Title: Evaluation of Safety and Efficacy of Intravenous Sulbactam-ETX2514 in the Treatment of Hospitalized Adults With Complicated Urinary Tract Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Entasis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS2514-2017-0003
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Results first posted 2019-06-05 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-06

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis
MeSH Terms: interventions — Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Intervention Model Description: This study is a double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of IV ETX2514SUL in patients with cUTIs.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulbactam-ETX2514 (ETX2514SUL) + Imipenem/Cilastatin (Experimental)
  Interventions: Drug: Sulbactam-ETX2514; Drug: Imipenem-cilastatin
- Placebo + Imipenem/Cilastatin (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Imipenem-cilastatin

INTERVENTIONS:
Drug: Sulbactam-ETX2514 — The ETX2514SUL regimen of 1 g ETX2514/1 g sulbactam infused over 3 hours q6h.
  Other Names: ETX2514SUL
  Arms: Sulbactam-ETX2514 (ETX2514SUL) + Imipenem/Cilastatin
Drug: Placebo — Matching 1g IV solution.
  Arms: Placebo + Imipenem/Cilastatin
Drug: Imipenem-cilastatin — All patients will receive background therapy with 500 mg IV imipenem/cilastatin q6h.

SUMMARY:
This study is a double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of IV ETX2514SUL in patients with complicated urinary tract infections (cUTIs) who are otherwise relatively healthy.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of IV ETX2514SUL in patients with cUTIs who are otherwise relatively healthy. Patients with Acute Pyelonephritis may also be enrolled. Approximately 80 patients will be randomized to receive either 1 g ETX2514/1 g sulbactam IV or matching placebo every 6 hours (q6h). All patients will receive background therapy with 500 mg IV imipenem/cilastatin q6h.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent form (ICF). If a study patient is unable to provide informed consent due to their medical condition, the patient's legally authorized representative may consent on behalf of the study patient as permitted by local law and institutional Standard Operating Procedures.
* Male or female, 18 to 90 years of age, inclusive.
* Expectation, in the judgment of the Investigator, that the patient's cUTI would require initial hospitalization and treatment with IV antibiotics.
* Documented or suspected cUTI or Acute pyelonephritis (AP).

Exclusion Criteria:

* Gross hematuria requiring intervention other than administration of study drug or removal or exchange of a urinary catheter.
* Known non-renal source of infection such as endocarditis, osteomyelitis, abscess, meningitis, or pneumonia diagnosed within 7 days prior to randomization that would interfere with evaluation of response to the study antibiotics.
* Patient requires continuing treatment with probenecid, methotrexate, ganciclovir, valproic acid, or divalproex sodium during the study.
* Receipt of a single dose of a long-acting, potentially-effective systemic antibiotic with activity against Gram-negative uropathogens for more than 24 hours within the 72-hour window prior to randomization.
* Requirement at time of randomization for any reason for additional systemic antimicrobial therapy (including antibacterial, antimycobacterial, or antifungal therapy) other than study drug, with the exception of a single oral dose of any antifungal treatment for vaginal candidiasis.
* Likely to require the use of an antibiotic for cUTI or AP prophylaxis during the patient's participation in the study [from randomization through the Late Follow-up (LFU) Visit].
* Any patients previously randomized in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anibal Calmaggi, MD, Study Chair — Medpace, Inc.
Locations (4):
- Bulgaria (4):
  - Universeity Multiprofile Hospital for Active Teatment, Sofia
  - University Multiprofile Hospital for Active Teatment-Clinic of Nephrology, Sofia
  - Multiprofile Hospital for Active Teatment (MHAT) and Emergency Medicine - Pirogov, Sofia
  - Multiprofile Hospital for Active Teatment (MHAT) and Emergency Medicine - Doverie, Sofia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sagan O, Yakubsevitch R, Yanev K, Fomkin R, Stone E, Hines D, O'Donnell J, Miller A, Isaacs R, Srinivasan S. Pharmacokinetics and Tolerability of Intravenous Sulbactam-Durlobactam with Imipenem-Cilastatin in Hospitalized Adults with Complicated Urinary Tract Infections, Including Acute Pyelonephritis. Antimicrob Agents Chemother. 2020 Feb 21;64(3):e01506-19. doi: 10.1128/AAC.01506-19. Print 2020 Feb 21. PMID 31843995

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sulbactam-ETX2514 (ETX2514SUL) + Imipenem/Cilastatin | Placebo + Imipenem/Cilastatin
Started | 53 | 27
Completed | 51 | 27
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulbactam-ETX2514 (ETX2514SUL) + Imipenem/Cilastatin | Placebo + Imipenem/Cilastatin | Total
Number analyzed (Participants) | 53 | 27 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (17.55) | 54.9 (15.92) | 52.6 (17.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 11 | 38
  Male | 26 | 16 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 52 | 27 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 53 | 27 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI (Body Mass Index) [Mean (Standard Deviation); unit: Kg/m^2] | 28.09 (6.661) | 28.63 (5.856) | 28.27 (6.368)
Height [Mean (Standard Deviation); unit: Centimeters] | 172.6 (8.81) | 173.1 (8.44) | 172.8 (8.63)
Weight [Mean (Standard Deviation); unit: Kilograms] | 83.79 (20.644) | 85.76 (17.929) | 84.45 (19.677)
Screening Creatinine Clearance [Mean (Standard Deviation); unit: Milliliters per minute] | 94.3 (23.76) | 91.7 (18.19) | 93.4 (21.96)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Success
Description: The primary efficacy endpoint for this study was the proportion of patients with an overall success (clinical cure and micro-biologic eradication) for the m-MITT (Micro-biologically Modified Intent-to-Treat) Population at the TOC Visit.
Time Frame: From baseline through day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Sulbactam-ETX2514 (ETX2514SUL) + Imipenem/Cilastatin | Placebo + Imipenem/Cilastatin
Number analyzed (Participants) | 47 | 21
Participants | 36 | 17

2. Secondary Outcome: Clinical Cure
Description: Proportion of patients with a response of clinical cure for the MITT(modified intent to treat), m-MITT (microbiologically modified intent to treat), CE(clinically evaluable), and ME(microbiologically evaluable) populations at the TOC(test of cure) visit.
Time Frame: Baseline to day 21
Population: The number analyzed for each population is different as the efficacy outcome is for the proportion of subjects with a clinical cure for each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Sulbactam-ETX2514 (ETX2514SUL) + Imipenem/Cilastatin | Placebo + Imipenem/Cilastatin
Number analyzed (Participants) | 53 | 27
Participants
  MITT population | 52 | 27
  m-MITT population: number analyzed (Participants) | 47 | 21
  m-MITT population | 46 | 21
  CE population: number analyzed (Participants) | 52 | 27
  CE population | 52 | 27
  ME population: number analyzed (Participants) | 45 | 21
  ME population | 45 | 21

3. Secondary Outcome: Microbiologic Eradication
Description: Proportion of patients with a response of microbiologic eradication for the m-MITT(microbiologically modified intent to treat) and ME(microbiologically evaluable) populations at the TOC visit
Time Frame: Baseline to day 21
Population: The analysis population differs for each group because the efficacy endpoint is for specific populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Sulbactam-ETX2514 (ETX2514SUL) + Imipenem/Cilastatin | Placebo + Imipenem/Cilastatin
Number analyzed (Participants) | 53 | 27
Participants
  m-MITT population: number analyzed (Participants) | 47 | 21
  m-MITT population | 37 | 17
  ME population: number analyzed (Participants) | 45 | 21
  ME population | 36 | 17

ADVERSE EVENTS:
Time Frame: 48 hours to day 1, day 1, day 2, day 3, day 4, day 5, day 6,Day 7 to 14/ EOT + 1 day, 7 days post-EOT +/- 1 day(TOC), 7 days post-TOC +/- 2 days (LFU)
Arm/Group | Sulbactam-ETX2514 (ETX2514SUL) + Imipenem/Cilastatin | Placebo + Imipenem/Cilastatin
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/27
Other Adverse Events (participants affected / at risk) | 8/53 | 3/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulbactam-ETX2514 (ETX2514SUL) + Imipenem/Cilastatin (N=53) | Placebo + Imipenem/Cilastatin (N=27)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Phlebitis (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03445195/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT03445195/SAP_001.pdf